CLINICAL TRIAL: NCT03051464
Title: A Phase III Study Testing Two Dose Escalation Strategies to Increase the Population of Complete Responders After Radiation Therapy in the Context of Organ Preservation for Patients With Rectal Cancer
Brief Title: No Surgery Trial / Two Dose-escalation Strategies
Acronym: Morpheus
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Te Vuong, Director, Radiation Oncology Department, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-301
Record Dates: First submitted 2017-02-07; First posted 2017-02-13 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Stage II Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemoradiation + EBRT Boost (Experimental): standard chemoradiation (45 Gy in 25 with concomitant 5-FU or Xeloda chemotherapy) and an external beam boost of 9 Gy in 5; Complete responders and Non-complete responders
  Interventions: Procedure: Complete responders and Non-complete responders; Radiation: Chemoradiation + EBRT Boost
- Chemoradiation + HDRBT Boost (Experimental): standard chemoradiation (45 Gy in 25 with concomitant 5-FU or Xeloda chemotherapy) and followed by a brachytherapy boost of 30 Gy in 3 fractions; Complete responders and Non-complete responders
  Interventions: Procedure: Complete responders and Non-complete responders; Radiation: Chemoradiation + HDRBT Boost

INTERVENTIONS:
Procedure: Complete responders and Non-complete responders — Patients that are complete responders will not have surgery. Patients that are non-complete responders will have surgery.
Radiation: Chemoradiation + EBRT Boost — 45 Gy in 25 with concomitant 5-FU or Xeloda chemotherapy) and an external beam boost of 9 Gy in 5
  Arms: Chemoradiation + EBRT Boost
Radiation: Chemoradiation + HDRBT Boost — 45 Gy in 25 with concomitant 5-FU or Xeloda chemotherapy) and followed by a brachytherapy boost of 30 Gy in 3 fractions
  Arms: Chemoradiation + HDRBT Boost

SUMMARY:
A randomized study of 131 patients. Patients with a clinical T2-3 N0 rectal cancer will be randomized to two arms (arm A: standard chemoradiation (45 Gy in 25 with concomitant 5-FU or Xeloda chemotherapy) and an external beam boost of 9 Gy compared to arm B: standard chemoradiation (45 Gy in 25 with concomitant 5-FU or Xeloda chemotherapy) and followed by a brachytherapy boost of 30 Gy in 3 fractions).

DETAILED DESCRIPTION:
It is becoming clear that there is a now an international consensus that rectal cancer research efforts need to be more focused in optimizing a non-surgical approach. This concept is very relevant to an ageing patient population with multiple co-morbidities regularly seen at the Jewish General Hospital and across the province. After interim analysis on 40 patients of the pilot study a phase III study is proposed. We are therefore proposing a phase III multicentric study of 145 patients to compare the two best known radiation dose escalation strategies and to achieve a complete clinical response. Patients with a clinical T2-3 N0-1 rectal cancer will be randomized to two arms (arm A: standard chemoradiation (45 Gy in 25 with concomitant 5-FU or Xeloda chemotherapy) and an external beam boost of 9 Gy compared to arm B: standard chemoradiation (45 Gy in 25 with concomitant 5-FU or Xeloda chemotherapy) and followed by a brachytherapy boost of 30 Gy in 3 fractions). Patients that have a high risk of recurrence or with more advanced stages of the disease will be excluded from the study, as only the local disease is being treated. The primary outcome for this proposal is rectum preservation in treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer patients, clinically staged as T2-T3 by MRI or endoscopic/trans-rectal ultrasound
* Rectal cancer staged as N0 by MRI or EUS/TRUS
* No metastatic lesion
* Rectal tumor occupying less than half of the circumference
* Tumor less than 5 cm on its largest dimension
* Tumor located at less than 10 cm from the anal verge
* Tumor penetration less than 5 mm in the mesorectal fat
* Tumor accessible for brachytherapy
* Lumen accessible for colonoscopy
* Patient should be a suitable candidate for brachytherapy and chemotherapy
* Older than 18 years of age
* Adequate birth control measures in women of childbearing potential
* Written informed consent

Exclusion Criteria:

* Patients with previous pelvic radiation
* Evidence of distant metastasis
* Extension of malignant disease to the anal canal
* Tumors staged as T4
* Tumors larger than 5 cm in length

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Estimated)
Dates: Start 2017-04-25 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
TME-free survival | 2 years post treatment
  Time from date of randomization to either TME or death in the intention to treat population

SECONDARY OUTCOMES:
Local Recurrence | 2 years post treatment
  Number of participants with Local recurrence as assessed by tests during follow-up visits.
Disease-free survival | 5 years post treatment
  The time between the date of randomization and recurrence, either in the pelvis or metastases. Patients without an event will be censored at the last date the patient was known to be disease-free.
Overall survival | 5 years post treatment
  The time between date of randomization and date of death due to any causes.
Overall Quality of life | 5 years post treatment
  Quality of life Questionnaires over different time point

CONTACTS AND LOCATIONS:
Overall Officials: Te Vuong, MD, Principal Investigator — Sir Mortimer Jewish General Hospital
Locations (4):
- Canada (4):
  - Hôpital Pierre Boucher, Longueuil, Quebec
  - Le Centre Hospitalier de l'Université de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Centre hospitalier universitaire de Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No